CLINICAL TRIAL: NCT01149668
Title: A Long-term Safety Study of the Pan-histone Deacetylase (HDAC) Inhibitor, PCI-24781, in Subjects With Cancer
Brief Title: A Safety and Tolerability Study of PCI-24781 in Subjects With Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pharmacyclics LLC. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCYC-0405-CA; PCI-24781 (Registry Identifier: 69451)
Record Dates: First submitted 2010-06-21; First posted 2010-06-23 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Lymphoma; Non-Hodgkin's Lymphoma; Hodgkin Disease; Multiple Myeloma; Leukemia; Lymphocytic
Keywords: PCI-24781; Lymphoma; Non-Hodgkin's; Hodgkin Disease; Multiple Myeloma; Leukemia; Lymphocytic; Chronic
MeSH Terms: conditions — Lymphoma; Lymphoma, Non-Hodgkin; Hodgkin Disease; Multiple Myeloma; Leukemia; Bronchiolitis Obliterans Syndrome | interventions — abexinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PCI-24781 (Experimental)
  Interventions: Drug: PCI-24781

INTERVENTIONS:
Drug: PCI-24781 — Subjects enrolled in this study will receive PCI-24781 administered orally at the schedule and dosage from their prior protocol.

SUMMARY:
The purpose of this study is to determine the long-term (> 6 months) safety of PCI 24781 PO in subjects with lymphoma.

DETAILED DESCRIPTION:
An open-label, monotherapy, multicenter, extension study open to subjects who have derived benefit from PCI 24781 PO for at least 6 months and want to continue receiving study drug.

Subjects enrolled in this study will receive PCI-24781 at the schedule and dosage from their prior protocol. Treatment may be continued as long as there is no evidence of progressive disease or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women with cancer that did not progress while treated with PCI 24781 PO for at least 6 months and who want to continue receiving study drug
2. Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2
3. Agreement to use contraception during the study and for 30 days after the last dose of study drug if sexually active and able to bear children
4. Willing and able to participate in all required evaluations and procedures in this study protocol including swallowing capsules without difficulty
5. Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information (in accordance with national and local subject privacy regulations)

Exclusion Criteria:

1. A life-threatening illness, medical condition or organ system dysfunction which, in the investigator's opinion, could compromise the subject's safety, interfere with the absorption or metabolism of oral PCI-24781, or put the study outcomes at undue risk
2. Significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of screening, or any Class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification
3. Malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel or ulcerative colitis, symptomatic inflammatory bowel disease, or partial or complete bowel obstruction
4. Immunotherapy, chemotherapy, radiotherapy, corticosteroids (at dosages equivalent to prednisone > 20 mg/day) or experimental therapy (other than PCI-24781 PO) within 4 weeks before first dose of study drug
5. Concomitant use of medicines known to cause QT prolongation or torsades de points (see Appendix 2)
6. Central nervous system involvement by lymphoma
7. Known history of Human Immunodeficiency Virus (HIV) or active infection with Hepatitis C Virus (HCV) or Hepatitis B Virus (HBV) or any uncontrolled active systemic infection
8. Creatinine > 1.5 x institutional upper limit of normal (ULN); total bilirubin > 1.5 x ULN (unless due to Gilbert's disease); and aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 2.5 x ULN
9. Lactating or pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2010-06; Primary Completion 2012-12 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Safety | 30 days after last dose of study drug
  frequency, severity and relatedness of adverse events

SECONDARY OUTCOMES:
Tumor Response | frequency of tumor assessments done per standard of care
  tumor response will be assessed per established response criteria. This study will capture time to disease progression and duration of response.

CONTACTS AND LOCATIONS:
Overall Officials: Thorsten Graef, MD, Study Director — Pharmacyclics LLC.
Locations (5):
- United States (5):
  - Northwestern Univ. Med School, Chicago, Illinois
  - Horizon Oncology Center, Lafayette, Indiana
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Univ. of Nebraska Medical Center, Omaha, Nebraska
  - Sarah Cannon Research Institute, Nashville, Tennessee